CLINICAL TRIAL: NCT05016336
Title: Strategy Based Cognitive Training Effects on Cognitive Performance of Older Adults in a Socially Interactive Learning Group
Brief Title: Cognitive Training and Social Interaction Effects on Cognitive Performance of Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bar-Ilan University, Israel (Other)
Responsible Party: Principal Investigator, Michal Lavidor, Principal Investigator, Bar-Ilan University, Israel
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 08082021ML
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Cognitive Decline
Keywords: Cognitive training; Strategy training; Older adults; Mnemonic; Social interaction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The study included 32 subjects, 20 in the experimental group and 12 in the control group. The experimental group received 12 sessions of strategy-based cognitive training combined with a socially interactive learning method. The control group received the same number of meetings but without the strategy training. Participants were recruited from designated active groups in the community.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- strategy-based cognitive training + social interaction (Experimental): The experimental group received twelve 60 minutes sessions of strategy-based cognitive training. (i.e., training in mnemonic memory strategies). We chose to train multiple strategies instead of a single one in effort to reach larger training gains. each session began with engaging conversations between the researcher and participants. After each practice trial, participants were encouraged to share their ideas/stories/associations or visual images (mnemonic uses) in turn. All other participants were allowed to give feedback relating to what can be learned from each mnemonic use or give their own ideas on how they think it can be improved.
  Interventions: Other: Social interaction combined with cognitive training based on mnemonic strategies.
- social interaction (Active Comparator): The social interaction control group received the same number of group meetings but without the strategy training. Meetings content consisted of providing tools for making social connections, providing tools for interpersonal communication and raising the participant's sense of personal well-being through group contact.
  Interventions: Other: Social interaction group

INTERVENTIONS:
Other: Social interaction combined with cognitive training based on mnemonic strategies. — In the first six sessions, participants in the experimental group learned and practiced six different mnemonic strategies: Story-Formation strategy, Face-Name strategy, Peg-Word strategy, Chunking strategy, Key-Word strategy and the Method of Loci. In the following six sessions, in order to assimilate the strategies they learned, participants practiced the same tasks.
  Arms: strategy-based cognitive training + social interaction
Other: Social interaction group — In the control group, each session also began with a conversation between the participants. The sessions then dealt with the content of interpersonal communication and the acquisition of tools for creating interpersonal relationships. Participants were asked to share the way they used the tools they acquired between sessions and received feedback from the other participants
  Arms: social interaction

SUMMARY:
Aging is associated with a decline in almost all aspects of cognitive functions, particularly memory. Recent research suggests that combining cognitive training with ongoing social interaction may aid in improving cognitive functioning for older adults. Furthermore, accumulative evidence suggests that strategy-based cognitive training may also improve the trainee's memory. In this study, the investigators examined the effects of a combined strategy-based cognitive training and a socially interactive learning method on cognitive performance and transfer effects in older adults.

DETAILED DESCRIPTION:
A major concern with the aging of the world's population is a higher prevalence of age-related impairment of cognitive functions. This concern highlights the need to identify quick and effective interventions that can preserve cognitive functions.

A growing body of literature supports the notion that cognitive training may assist in promoting healthy brain aging and improve a wide range of cognitive abilities.

Cognitive training refers to a protocol consisting of a set of exercises designed to improve performance in one or several cognitive abilities. One approach to cognitive training mentioned in the literature is strategy training. Strategy training usually focuses on teaching specific strategies designed to help encode or retrieve information and involves techniques such as rehearsal, chunking, mental imagery, and story-formation.

A possible means for improving cognitive training outcomes is employing a socially interactive group-based cognitive training program versus an individual one. An abundance of studies has shown that social interaction may contribute to the slowing down of cognitive decline in old age.

Recent studies suggest that social interaction alone may not be beneficial for enhancing cognitive abilities, but when combined with a mental stimulus that requires cognitive effort, such improvement might be achieved.

Only a few studies to date have investigated the advantage of strategy training performed in-group vs individually and even fewer studies focused specifically on socially interactive learning methods. A recent pilot study combined cognitive training with social interaction for people with mild to moderate dementia and reported a significant cognitive improvement in favor of the social interaction group compared to the control group who was engaged in cognitive training only.

Social cognition is supported by an extensive system of limbic, cortical and subcortical brain regions. Many of these regions are also involved in episodic memory, semantic memory and other cognitive functions. Thus, it is possible that aspects of cognitive processing, which are activated through social interaction will also strengthen these cognitive abilities.

Engaging in social interaction usually consists of complex cognitive and memory challenges, which in turn may aid in enhancing cognitive abilities and cognitive reserve Training in a group setting can provide participants with an opportunity to problem-solve with a relevant peer group and allow individuals to gain comfort from sharing their concerns about memory.

The purpose of the current study was therefore to determine the effectiveness of a strategy-based cognitive training approach combined with a socially interactive learning method on cognitive performance and transferability of training gains for older adults.

Procedure:

Meetings of both groups were held in public community centers. A pre-session meeting was devoted to explaining the research objectives and signing consent forms. Prior to the first training meeting and after the program ended, cognitive evaluation measurements were taken individually from each subject. Before the final cognitive evaluation, participants were reminded to use the learned strategies.

Sample size assessment:

A priori power analysis using pilot data and the SimR package in R (version 1.0.5) suggested that 30 participants would provide sufficient power (power > 80%) to detect the critical strategy training plus social interaction effect on cognitive performance.

Statistical analysis plan:

Data will be analyzed with IBM SPSS Statistics for Windows, version 23 (IBM Corp., Armonk, N.Y., USA). The main analysis 'שד a mixed-design analysis that compares the experimental conditions (between-subject factors) regarding their effect on cognitive performance in 4 cognitive tests and 2-time points (within-subjects variables).

ELIGIBILITY:
Inclusion Criteria:

• Healthy participants who are active in a designated group in the community.

Exclusion Criteria:

• Any diagnosis of cognitive decline.

Min Age: 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2019-02-03 (Actual); Study Completion 2019-02-24 (Actual)

PRIMARY OUTCOMES:
Verbal Fluency Test (Chiu et al., 1997) | Change from baseline (before treatment) to immediately after treatment (12 weeks)
  Participants were asked to say aloud as many words as possible belonging to a given category (animal's category and fruit and vegetables category) within a period of sixty seconds.

SECONDARY OUTCOMES:
Wechsler Digit Span Test (Wechsler 2008) | Change from baseline (before treatment) to immediately after treatment (12 weeks)
  Series of digits were presented verbally at a rate of one digit per second. Subjects were required to repeat the digits verbally in the order presented.
Words Recall Test (Fairchild et al., 2013) | Change from baseline (before treatment) to immediately after treatment (12 weeks)
  Subjects were asked to remember a list of 16 words and to recall the list after a 5-min delay.
Corsi Block-Tapping Test (Corsi 1972) | Change from baseline (before treatment) to immediately after treatment (12 weeks)
  The task involves mimicking the researcher as he taps a sequence of up to nine identical spatially separated blocks.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Lavidor, Prof., Principal Investigator — Department of Psychology, and the Gonda Brain Research center, Bar Ilan University
Locations (1):
- Bar Ilan University, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analyzed during the current study are available from the main author.

REFERENCES:
- [Result] Choi M. Association between social participation and cognitive function among community-dwelling older adults living alone: Analysis of a nationally representative survey. Int J Nurs Pract. 2020 Aug;26(4):e12841. doi: 10.1111/ijn.12841. Epub 2020 May 27. PMID 32458529
- [Result] Hikichi H, Kondo K, Takeda T, Kawachi I. Social interaction and cognitive decline: Results of a 7-year community intervention. Alzheimers Dement (N Y). 2016 Dec 21;3(1):23-32. doi: 10.1016/j.trci.2016.11.003. eCollection 2017 Jan. PMID 29067317
- [Result] Krueger KR, Wilson RS, Kamenetsky JM, Barnes LL, Bienias JL, Bennett DA. Social engagement and cognitive function in old age. Exp Aging Res. 2009 Jan-Mar;35(1):45-60. doi: 10.1080/03610730802545028. PMID 19173101
- [Result] Park DC, Gutchess AH, Meade ML, Stine-Morrow EA. Improving cognitive function in older adults: nontraditional approaches. J Gerontol B Psychol Sci Soc Sci. 2007 Jun;62 Spec No 1:45-52. doi: 10.1093/geronb/62.special_issue_1.45. PMID 17565164
- [Result] Chan MY, Haber S, Drew LM, Park DC. Training Older Adults to Use Tablet Computers: Does It Enhance Cognitive Function? Gerontologist. 2016 Jun;56(3):475-84. doi: 10.1093/geront/gnu057. Epub 2014 Jun 13. PMID 24928557
- [Result] Iizuka A, Suzuki H, Ogawa S, Kobayashi-Cuya KE, Kobayashi M, Inagaki H, Sugiyama M, Awata S, Takebayashi T, Fujiwara Y. Does social interaction influence the effect of cognitive intervention program? A randomized controlled trial using Go game. Int J Geriatr Psychiatry. 2019 Feb;34(2):324-332. doi: 10.1002/gps.5024. Epub 2018 Dec 10. PMID 30430635
- [Result] Myhre JW, Mehl MR, Glisky EL. Cognitive Benefits of Online Social Networking for Healthy Older Adults. J Gerontol B Psychol Sci Soc Sci. 2017 Sep 1;72(5):752-760. doi: 10.1093/geronb/gbw025. PMID 26984523
- [Result] Cavallini E, Dunlosky J, Bottiroli S, Hertzog C, Vecchi T. Promoting transfer in memory training for older adults. Aging Clin Exp Res. 2010 Aug;22(4):314-23. doi: 10.3275/6704. Epub 2009 Nov 27. PMID 19966535
- [Result] Valentijn SA, van Hooren SA, Bosma H, Touw DM, Jolles J, van Boxtel MP, Ponds RW. The effect of two types of memory training on subjective and objective memory performance in healthy individuals aged 55 years and older: a randomized controlled trial. Patient Educ Couns. 2005 Apr;57(1):106-14. doi: 10.1016/j.pec.2004.05.002. PMID 15797159
- [Result] Rouse HJ, Small BJ, Faust ME. Assessment of Cognitive Training & Social Interaction in People with Mild to Moderate Dementia: A Pilot Study. Clin Gerontol. 2019 Jul-Sep;42(4):421-434. doi: 10.1080/07317115.2019.1590489. Epub 2019 Mar 21. PMID 30895883
- [Result] Bennett DA, Schneider JA, Tang Y, Arnold SE, Wilson RS. The effect of social networks on the relation between Alzheimer's disease pathology and level of cognitive function in old people: a longitudinal cohort study. Lancet Neurol. 2006 May;5(5):406-12. doi: 10.1016/S1474-4422(06)70417-3. PMID 16632311
- [Result] Ertel KA, Glymour MM, Berkman LF. Effects of social integration on preserving memory function in a nationally representative US elderly population. Am J Public Health. 2008 Jul;98(7):1215-20. doi: 10.2105/AJPH.2007.113654. Epub 2008 May 29. PMID 18511736
- [Result] Verhaeghen P, Marcoen A, Goossens L. Improving memory performance in the aged through mnemonic training: a meta-analytic study. Psychol Aging. 1992 Jun;7(2):242-51. doi: 10.1037//0882-7974.7.2.242. PMID 1535198
- [Result] Flynn TM, Storandt M. Supplemental group discussions in memory training for older adults. Psychol Aging. 1990 Jun;5(2):178-81. doi: 10.1037//0882-7974.5.2.178. PMID 2378683
- [Result] Chiu HF, Chan CK, Lam LC, Ng KO, Li SW, Wong M, Chan WF. The modified Fuld Verbal Fluency Test: a validation study in Hong Kong. J Gerontol B Psychol Sci Soc Sci. 1997 Sep;52(5):P247-50. doi: 10.1093/geronb/52b.5.p247. PMID 9310094
- [Result] Fairchild JK, Friedman L, Rosen AC, Yesavage JA. Which older adults maintain benefit from cognitive training? Use of signal detection methods to identify long-term treatment gains. Int Psychogeriatr. 2013 Apr;25(4):607-16. doi: 10.1017/S1041610212002049. Epub 2012 Dec 14. PMID 23237099
- [Result] Wechsler, D. (2008). Wechsler Adult Intelligence Scale-Fourth Edition: Administration and Scoring Manual. San Antonio, TX: Pearson Assessment.
- [Result] Corsi, P. M. (1972). Human memory and the medial temporal region of the brain.